CLINICAL TRIAL: NCT00997919
Title: A Phase I, Single-Dose, Randomized, Parallel-Group, Open-Label Study of the Safety, Tolerability, Pharmacokinetics, and Bioavailability of IV and SC MABT5102A in Healthy Volunteers
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics, and Bioavailability of IV and SC MABT5102A in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABE4662g
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — crenezumab

ARMS (2):
- A (Experimental)
  Interventions: Drug: MABT5102A
- B (Experimental)
  Interventions: Drug: MABT5102A

INTERVENTIONS:
Drug: MABT5102A — single SC dose
  Arms: A
Drug: MABT5102A — single IV dose
  Arms: B

SUMMARY:
This Phase I, single-dose, randomized, parallel-group, open-label study will evaluate the safety, tolerability, and pharmacokinetics of MABT5102A following subcutaneous (SC) and intravenous (IV) administration in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria

* Male subjects aged 18-50 years and female subjects aged 18-50 years who are not of childbearing potential and who are in good general health at the screening visit
* Body weight between 50 and 100 kg
* For male subjects of reproductive potential, a reliable means of contraception must be used (e.g., abstinence or a condom) for the duration of the study

Exclusion Criteria

* Female subjects with reproductive potential.
* Subjects with evidence of clinically significant neurologic, psychiatric, hepatic, renal, hematologic, pulmonary, respiratory, immunologic system abnormalities, acute infection, or other unstable medical disease
* Subjects with any malignancy (with the exception of completely excised basal cell or squamous cell carcinoma of the skin)
* History of alcohol, drug, or substance abuse within 6 months prior to randomization that, in the judgment of the investigator, may put the subject at risk for being unable to participate fully in the study for the duration of the study
* Past history of seizures, with the exception of childhood febrile seizures
* Clinically significant laboratory or ECG abnormalities
* Hospitalization during the 4 weeks prior to screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events, laboratory abnormalities, physical and neurological examination findings, vital signs, electrocardiogram (ECG) results) | Until study discontinuation

SECONDARY OUTCOMES:
Pharmacokinetic/Pharmacodynamic (area under the concentration-time curve, volume of distribution, clearance [CL] and apparent CL, terminal half-life) | Until study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Robert Paul, Ph.D., M.D., Study Director — Genentech, Inc.